CLINICAL TRIAL: NCT02409199
Title: A Randomized, Multicenter Study To Evaluate The Efficacy And Safety Of Apatinib Versus Docetaxel In Patients With Previously Treated Locally Advanced Or Metastatic Gastric Cancer, Including Adenocarcinoma Of The Gastroesophageal Junction
Brief Title: A Study of Apatinib Versus Docetaxol Patients With Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Tianshu Liu, Medicine-Oncology Derpartment of Zhongshan hospital, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-G301
Record Dates: First submitted 2015-03-26; First posted 2015-04-06 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Gastric Carcinoma
Keywords: Gastric Carcinoma; apatinib
MeSH Terms: conditions — Stomach Neoplasms | interventions — Docetaxel; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- apatinib (Experimental): Apatinib 850 mg qd po, and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: apatinib
- Docetaxel (Active Comparator): Docetaxel 60mg/m2 ivgtt every 3 weeks, and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel
  Arms: Docetaxel
Drug: apatinib
  Arms: apatinib

SUMMARY:
This multicenter, randomized study will evaluate the efficacy and safety of apatinib compared to docetaxel treatment in patients with advanced gastric cancer. At the start of the trial, patients will be randomized to one treatment arm: Arm A: apatinib 850mg qd every 3 weeks; Arm B: docetaxel 60mg/m2 every 3 weeks. Tumor assessment will be done every 8 weeks according to RECIST 1.1. The primary endpoint is progression free survival (PFS).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, aged ≥18 years;
* Histologically confirmed advanced or metastatic adenocarcinoma of gastric cancer(AGC) , including adenocarcinoma of the gastroesophageal junction ;
* At least one measurable and evaluable disease based on response evaluation criteria in solid tumors (RECIST v1.1);
* Patients must have received one prior chemotherapy regimen for AGC;First-line therapy must have included a combination of at least a platinum-based treatment given concurrently, and must have experienced disease progression during or after first-line therapy for their disease;
* Eastern Cooperative Oncology Group(ECOG) performance status of 0 or 1;
* Life expectancy of more than 3 months;
* Duration from the last therapy is more than 6 weeks for nitroso or mitomycin, More than 4 weeks for other cytotoxic agents, operation or radiotherapy;
* Adequate hepatic, renal, heart, and hematologic functions ( hemoglobin≥ 90g/L, platelets ≥ 80 × 109/L, neutrophil ≥1.5 × 109/L, serum creatinine≤ 1.5mg/dl, total bilirubin ≤1.5 ×ULN, and serum transaminase≤2.5×ULN);

Exclusion Criteria:

* Pregnant or lactating women;
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma insitu of uterine cervix;
* Prior chemotherapy regimen have included taxane (docetaxel or paclitaxel); Uncontrolled hypertension;
* Intercurrence with one of the following: coronary artery disease, arrhythmia and heart failure;
* Urine protein>grade 1;
* Any factors that influence the usage of oral administration;
* patients with a clear tendency of gastrointestinal bleeding;
* Abnormal coagulation function(INR≥1.5, APTT≥1.5 ULN);
* Abuse of alcohol or drugs;
* Less than 4 weeks from the last clinical trial;
* Prior treatment with antivascular endothelial growth factor or the other anti angiogenesis therapy;
* Evidence of central nervous system(CNS) metastasis;
* Disability of serious uncontrolled intercurrence infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Approximately 1 year
  defined as the time from randomize to progression or death; RECIST guidelines were used to define all responses after patients had received every 8 weeks of therapy

SECONDARY OUTCOMES:
Overall survival (OS) | Approximately 3 years
  defined as the time from randomize to death
Objective response rate (ORR) | Approximately 1 year
  defined as the rate of complete response and partial response according to RECIST guidelines.
Disease control rate(DCR) | Approximately 1 year
  defined as the rate of complete response , partial response and stable disease according to RECIST guidelines.
Quality of life(QoL) | Approximately 3 years
  as measured by the European Organization for Research and Treatment of Cancer questionnaire (EORTC QLQ C30)
Safety (incidence of adverse events) | Approximately 1 year
  incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Liu Tianshu, doctor, Principal Investigator — oncology department
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China